CLINICAL TRIAL: NCT01462396
Title: Phase I Study of Allogeneic Stem Cell Transplantation for Advanced Neuroblastoma Using Major Histocompatibility Complex (MHC) Mismatched Related Donors and Sub-Myeloablative Regimen
Brief Title: Allogeneic Stem Cell Transplantation for Advanced Neuroblastoma Using MHC Mismatched Related Donors
Acronym: STALLO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Principal Investigator, Doug Myers, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STALLO
Record Dates: First submitted 2011-10-25; First posted 2011-10-31 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Relapsed; Refractory
MeSH Terms: conditions — Neuroblastoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Haploidentical allogeneic stem cell transplant following sub-myeloablative conditioning and cell selection using the Miltenyi Clinimacs device
  Interventions: Device: CD34+ cells selected with the Miltenyi Clinimacs machine

INTERVENTIONS:
Device: CD34+ cells selected with the Miltenyi Clinimacs machine — Haploidentical allogeneic stem cell transplant following sub-myeloablative conditioning and cell selection using the Miltenyi Clinimacs device

SUMMARY:
Allogeneic stem cell transplantation has been explored for patients with high risk neuroblastoma. Results have been mixed, with only small series and case reports. Recent reports, however, especially with haploidentical transplantation have been more encouraging. Eradication of neuroblastoma may be mediated by both components of the innate immune system (natural killer cells) and through the adaptive immune system via T-cell cytotoxicity and the development of a humoral response to tumor specific antigens and minor histocompatibility antigens. To overcome restrictions created by unavailability of Human leukocyte antigen (HLA) matched donors, stem cell grafts from haploidentical related donors have been explored. Historically, the use of full haplotype mismatched family member donors has been limited by the development of severe graft-versus-host disease and the high rate of graft failure. Graft failure can now be overcome by increasing immunosuppression and increasing the number of transplanted stem cells. The most effective means of graft versus host disease (GVHD) prophylaxis is T cell depletion of the donor marrow. A 3-4 log depletion will reduce the risk of developing significant GVHD to less than 10%. Methods to mobilize stem cells from the bone marrow into the peripheral blood and collect these stem cells by apheresis now increase the availability of stem cells by a magnitude. Selection devices have been developed that will prepare extremely pure populations of these CD34 cells with upwards of 5 logs depletion of contaminating T cells. The CliniMACS CD34 Reagent System is a medical device designed to select CD34+ hematopoietic cells from heterogeneous hematologic cell populations. The investigators intend to provide mismatched related hematopoietic stem cell transplantation to up to 10 patients with relapsed refractory neuroblastoma. Harnessing the potential for innate and adaptive immune responses through allogeneic Hematopoietic stem cell transplantation (HSCT) may provide cure for some patients with this tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - <18 years
* Measurable tumor by routine imaging or bone marrow biopsy
* Patient must have an 3/6, 4/6, or 5/6 human leukocyte antigen (HLA)-mismatched related donor who is Epstein-Barr virus (EBV) seropositive
* Karnofsky score 60% or greater if 10yrs old or older, Lansky score 60% or greater if under 10yrs old
* Pulse ox >90% on room air
* Recovered from toxic effects of prior chemotherapy
* Patient must not be pregnant
* Patient must be HIV negative
* Patient or responsible person must be able to understand and sign an informed consent
* Available donor without contraindication for stem cell collection

Exclusion Criteria:

* Pregnant and lactating women.
* Human immunodeficiency virus (HIV) positive patient.
* Uncontrolled intercurrent infection.
* Renal failure (Creatine > 1.5 or Creatinine Clearance < 40 ml/min/1.73m2)
* Active hepatitis or cirrhosis with liver test values greater than 3 times normal
* NOTE: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion, after review by the Children's Mercy Hospital ethics board
* Donor Inclusion/Exclusion Criteria
* Donor must be in good health based on review of systems and results of physical examination, and routine testing per standards of good medical care.
* Female donors of childbearing age must have a negative pregnancy test and must not be lactating
* EBv seropositive
* Donor stem cells should be human leukocyte antigen (HLA) typed using molecular methods. See section 6.1.3 for HLA matching requirements.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The immediate safety of a fludarabine based reduced intensity conditioning regimen and CD34+ stem cell selected mis-matched, related, allogeneic transplant will be assess in patients with relapsed/refractory neuroblastoma | 6 weeks
  Monitoring of mortality, toxicity (NCI Common Criteria), acute and chronic graft versus host disease, engraftment rate will contribute to safety assessment

SECONDARY OUTCOMES:
Infusional and long term safety and persistence of tumor redirected, genetically modified, donor derived, allogeneic multi-virus specific cytotoxic T-cells (tV-CTL) after allogeneic hematopoietic stem cell transplant in patients with neuroblastoma | 4-8 weeks post transplant
  Tumor evaluation will occur 4-8 weeks after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Myers, MD, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Children's Mercy Hospital — http://www.childrensmercy.org/